CLINICAL TRIAL: NCT03154892
Title: The Effect of Conbercept Injection Through Different Routes for Neovascular Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Conbercept Injection
Record Dates: First submitted 2017-05-07; First posted 2017-05-16 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Neovascular Glaucoma
MeSH Terms: conditions — Glaucoma, Neovascular | interventions — Intracameral Injection; Intravitreal Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intracameral injection (Experimental): Intracameral injection of conbercept for the treatment of NVG
  Interventions: Procedure: Intracameral injection
- Intravitreal injection (Active Comparator): Intravitreal injection of conbercept for the treatment of NVG
  Interventions: Procedure: Intravitreal injection

INTERVENTIONS:
Procedure: Intracameral injection — Intracameral Conbercept injection for the treatment of NVG
  Arms: Intracameral injection
Procedure: Intravitreal injection — Intravitreal Conbercept injection for the treatment of NVG
  Arms: Intravitreal injection

SUMMARY:
The neovascular glaucoma (NVG) is a refractory type of secondary glaucoma and often lead to frustrated treatment and blindness. It has been confirmed high levels of vascular endothelial growth factor (VEGF) in NVG. Conbercept is an anti-VEGF agent，its role in regression of other neovascular disorders such as wet-type age-related macular degeneration and diabetic retinopathy has been described. Investigators aim to evaluate the efficacy and safety of intracameral and intravitreal injection of conbercept for the treatment of NVG.

DETAILED DESCRIPTION:
The neovascular glaucoma (NVG) is a refractory type of secondary glaucoma and often lead to frustrated treatment and blindness. It has been confirmed high levels of vascular endothelial growth factor (VEGF) in NVG. Conbercept is an anti-VEGF agent，Its role in regression of other neovascular disorders such as wet-type age-related macular degeneration and diabetic retinopathy has been described. The intravitreal injection of anti-VEGF agent has shown its therapeutic potential for the early stage of NVG, but not for the late stage. Intracameral injection maybe used as an alternative way for administration. Investigators aim to evaluate the efficacy and safety of intracameral and intravitreal injection of conbercept for the treatment of NVG.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of neovascular glaucoma (Stage 1-2-3)
* Individuals who are ages 20-80 years old; male or female of chinese
* Visual acuity of light perception or better in the study eye
* Willing and able to comply with clinic visits and study-related procedures
* Provide signed informed consent

Exclusion Criteria:

* Use of intraocular anti-VEGF agents in the study eye in the past 3 months.
* Active ocular or periocular infection in the study eye
* Uncontrolled Blood Pressure
* Thromboembolism
* Congestive Heart Failure
* Renal Failure
* History of myocardial infarction
* History of Stroke
* Pregnant or breast-feeding women
* Participation in another simultaneous medical investigator or trial

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
NVI/NVA | 1 week and 1 month after operation
  Changes in extent of iris or angle neovascularization

SECONDARY OUTCOMES:
IOP | 1 week and 1 month after operation
  Changes in Intraocular pressure
BCVA | 1 week and 1 month after operation
  Changes in best corrected visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Ling Bai, MD,PhD, Principal Investigator — Second affiliated hospital of Xian Jiaotong University
Locations (1):
- Department of Ophthalmology, Second affiliated hospital of Xian Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

REFERENCES:
- [Derived] Bai L, Wang Y, Liu X, Zheng Y, Wang W, He N, Tariq F, Wang F, Zhang S. The Optimization of an Anti-VEGF Therapeutic Regimen for Neovascular Glaucoma. Front Med (Lausanne). 2022 Jan 10;8:766032. doi: 10.3389/fmed.2021.766032. eCollection 2021. PMID 35083234